CLINICAL TRIAL: NCT03788499
Title: Randomized, Controlled Clinical Study of Using Massage of Maxillofacial and Oral Cavity to Prevent Oral Mucositis in Patients With Nasopharyngeal Carcinoma Undergoing Radiotherapy
Brief Title: Using Massage of Maxillofacial and Oral Cavity to Prevent Radioactive Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XQonc-009
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Massage; Maxillofacial and Oral Cavity; Radioactive Oral Mucositis; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): routine oral care and functional exercise.
- Massage arm (Experimental): Massage of Maxillofacial and oral cavity plus routine oral care and functional exercise
  Interventions: Other: Massage of Maxillofacial and Oral Cavity

INTERVENTIONS:
Other: Massage of Maxillofacial and Oral Cavity — Massage of Maxillofacial and Oral Cavity is performed five times a day, each part lasts 1-2 minutes, repeating 3 cycles. The maxillofacial and oral massage last from the first day of radiotherapy to three months after last radiotherapy.
  Arms: Massage arm

SUMMARY:
A total of 160 cases of nasopharyngeal carcinoma patients who met the inclusion criteria were randomly assigned to two groups. The experimental group was given massage of maxillofacial and oral cavity plus routine oral care and functional exercise. The control group was given routine oral care and functional exercise. Analyze the difference of incidence of severe acute radioactive oral mucositis in these two groups.

DETAILED DESCRIPTION:
160 nasopharyngeal carcinoma patients were enrolled and randomly assigned to two groups in a 1:1 ratio. The experimental group was given massage of maxillofacial and oral cavity plus routine oral care and functional exercise, the control group was only given routine oral care and functional exercise. Assess the condition of oral mucosa, according to the grading standard of RTOG acute radiation injury, everyday during radiotherapy. After radiotherapy, follow up the condition of oral mucosa one time per month for a total three times. Then analyze the incidence difference between two groups.

massage method：The duration of the massage lasts from the first day of radiotherapy to three months after the end of radiotherapy，5 times a day（After getting up, before breakfast, lunch, dinner and going to bed). massage of maxillofacial includes the left and right cheeks, the upper jaw, the lower jaw, and around the mouth. Oral Massage includes the tongue, hard palate, the gums, and the bucca. Each part lasts 1-2min，repeating 3 cycles each time. Patients who could finished at least 75% are included in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed by pathology with nasopharyngeal carcinoma;
2. ECOG PS: 0-2;
3. Gender is not limited, Age between 18 years old and 70 years old.
4. Clear consciousness, no mental illness or cognition impairment;
5. The expected survival time is more than 12 months;

Exclusion Criteria:

1. Patients with other severe diseases affecting the quality of life or the treatment process;
2. Unwilling to actively cooperate with investigators;
3. Patients with previous oral diseases;
4. Patients who have received head and neck surgery and radiotherapy;
5. A history of psychotropic substance abuse or a mental disorder;
6. Participated in clinical trials of other anti-tumor drugs within 4 weeks before enrollment;
7. Women who are pregnant or in lactation;
8. Other situations that may affect the results of the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of severe radioactive oral mucositis | 3 months
  the status of oral mucosa was evaluated daily during radiotherapy. According to the grading standard of RTOG acute radiation injury, statistical analysis was made on whether there was a difference and statistical significance in the incidence rate of oral mucositis with radiation above grade 3 between the two groups.

SECONDARY OUTCOMES:
the time at which the radioactive oral mucosa occurred; Difficulty in opening your mouth. | 3 months
  the time at which the radioactive oral mucosa occurred; Difficulty in opening your mouth.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality
  - the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality